CLINICAL TRIAL: NCT02654548
Title: Sebum Excretion in Neonates of Women With Polycystic Ovary Syndrome (PCOS): Does Increased Skin Greasiness in the First Week of Life Predict Subsequent Development of the Syndrome? A Cohort Study
Brief Title: Sebum Excretion in Neonates of Women With Polycystic Ovary Syndrome (PCOS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Homerton University Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FE1302
Record Dates: First submitted 2016-01-11; First posted 2016-01-13 (Estimated); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PCOS women and babies (Experimental): Sebum output using Sebutape on post-partum PCOS women and new born babies.
  Interventions: Other: Sebutape
- Non-PCOS women and babies (Active Comparator): Sebum output using Sebutape on post-partum non-PCOS women and new born babies.
  Interventions: Other: Sebutape

INTERVENTIONS:
Other: Sebutape — Women who consent to the study will have a sebutape attached to their and their babies foreheads to measure the levels of androgens.

SUMMARY:
To investigate whether women with polycystic ovary syndrome who are post-partum excrete higher levels of sebum in comparison to healthy controls due to high levels of androgens.

DETAILED DESCRIPTION:
First degree relatives of women with PCOS have a 3-4 fold increased prevalence of the syndrome compared with the general population, suggesting an inherited genetic predisposition. Many investigations into possible candidate genes for PCOS susceptibility have hypothesised the incomplete penetrance of a dominant gene, although no consensus has been achieved as to any exact genetic polymorphisms which may be culpable.

Primate studies have offered credence to the theory that genomic imprinting is influenced by environmental hyperandrogenism and the hypothesis of intra-uterine exposure to excess androgens as a cause of PCOS is gaining momentum (Abbott et al, 2010). At birth, both mother and neonate are influenced by an identical hormone profile, and it is therefore expected that sebum excretion rates (a correlate of androgen excess) will be higher in those neonates born to mothers with PCOS when compared to those without. This would account for the observed familial transition of PCOS (Legro et al, 1998; Vink et al, 2006), and support the hypothesis that in-utero hyperandrogenism primes differentiating tissues for later expression of the PCOS phenotype in adolescence.

ELIGIBILITY:
Inclusion Criteria:

* Women (with and without a diagnosis of polycystic ovarian syndrome) aged 18-40 with an uncomplicated singleton pregnancy, who deliver a female baby at term (37 weeks gestation or longer). Women in the PCOS cohort will be defined by all the ESHRE/ASRM Rotterdam criteria. Women in the control group, non-PCOS who deliver a female baby will be age matched to the PCOS group. Conception method (natural/assisted) and maternal parity does not affect inclusion but will be documented for subsequent analysis.

Exclusion Criteria:

* baby boys

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Sebum output using Sebutape | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Roy Homburg, FROG, Principal Investigator — Professor
Locations (1):
- Homerton Fertility Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Homburg R, Gudi A, Shah A, M Layton A. A novel method to demonstrate that pregnant women with polycystic ovary syndrome hyper-expose their fetus to androgens as a possible stepping stone for the developmental theory of PCOS. A pilot study. Reprod Biol Endocrinol. 2017 Aug 8;15(1):61. doi: 10.1186/s12958-017-0282-1. PMID 28789693